CLINICAL TRIAL: NCT02522442
Title: Phase IV Study of Bi-Level Positive Positive Airway Pressure (BiPAP)Compared to Nasal Continuous Positive Airway Pressure (CPAP) Therapy
Brief Title: Auto Bilevel Adherence Following a Poor Initial Encounter With Continuous Positive Airway Pressure (CPAP)
Acronym: BiPAPRescue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Collaborators: Mayo Clinic (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ABF-2007-MCT-03
Record Dates: First submitted 2011-07-18; First posted 2015-08-13 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Auto BiLevel Group (Experimental): Auto Bilevel; auto-titrating bilevel positive airway pressure device with pressure flexing used as experimental treatment for obstructive sleep apnea
  Interventions: Device: Auto BiLevel
- CPAP Group (Active Comparator): CPAP; continuous positive airway pressure used as comparator treatment for obstructive sleep apnea
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure
  Arms: CPAP Group
Device: Auto BiLevel — Auto Bilevel positive airway pressure with Flex
  Arms: Auto BiLevel Group

SUMMARY:
The primary objective outcome is the proportion of participants compliant (at least four hours of use per night for all nights) in the Auto Bilevel group compared to the continuous positive airway pressure (CPAP) group after 90 days of treatment during the investigation. Proportion will be calculated using the cumulative number of hours on therapy divided by the total number of days of the investigation for each participant. The mean and standard deviation of these mean therapy hours will then be calculated for each arm of the investigation. Participants with compliance of at least four hours will be classified as "compliant" and those with less than four hours will be classified as "non-compliant". The null hypothesis will be rejected if the mean of the primary objective outcome for all participants in the BiPAP® Auto with Bi-Flex® therapy (auto Bilevel) arm is significantly greater than that for all participants in the CPAP therapy arm

DETAILED DESCRIPTION:
Initial Screening

It is preferred that participant's are recruited the morning after their failed clinical CPAP titration in the lab. Participants are able to be enrolled within ninety days following this failure if circumstances preclude approach and consent the morning after titration failure. Participants will be asked to wear the Actiwatch for approximately seven days prior to the clinical titration polysomnogram (PSG; and again for seven days prior to their final visit .) Actiwatch is worn on the participant's wrist to assess sleep continuity. Participants will be asked to press the "Marker button" on the Actiwatch when they get in bed each night to have a documented time mark when the device is downloaded. Participants will also be asked to fill in the sleep diary (provided by sleep clinic) during the seven days (14 days total; 7 at the beginning of the study and 7 days prior to the 90 Day visit) they use the Actiwatch.

Randomization/Therapy Initiated (Visit #1)

Participants will be randomized and scheduled for a BiPAP® Auto with Bi-Flex® titration or CPAP titration night in the lab. General therapy titration guidelines are documented in Appendix I & II (see Appendix I & II at end of document). Heart Rate Variability (HRV) will be assessed at both the diagnostic portion and titration portion of the research PSG. During the diagnostic portion of the research PSG, HRV needs to be assessed for ten minutes while the participant is awake. At the end of the titration portion of the research PSG, the HRV needs to be assessed for ten consecutive minutes while the participant is awake.

Enrolled participants will then complete a questionnaire to assess functional outcomes of sleep quality (FOSQ), Epworth Sleepiness Scale (ESS), Visual Analog Scale (VAS) for mask comfort and satisfaction with therapy, Psychomotor Vigilance Task (PVT), attitudes toward use measurement, and Fatigue Severity Scale (FSS; see Appendix III for description of measurements).

Participants will be set up with their respective machines after titration or within ten days (10 +/- 2) days of titration and will take these devices home for the next three months. Thus, total participation in the trial will be on average 3-4 months. All positive airway pressure machines will include a programmed SmartCard to monitor objectively compliance. Participants randomized to standard CPAP therapy will receive a SmartCard programmed to provide CPAP at their prescribed pressure. Both the participant and the sleep health staff administering the questionnaires and psychomotor vigilance task, will be blinded to the therapy the SmartCard is programmed to provide. Participants randomized to novel therapy will receive a SmartCard programmed to provide BiPAP® Auto with Bi-Flex®. The SmartCard programming will be done by an unblinded study staff member. The settings for the novel therapy will be:

* Min Expiratory Positive Airway Pressure (EPAP) = 4 cmH2O for prescribed CPAP ≤ 10 cmH2O (use 6 cmH2O for prescribed CPAP > 10 cmH2O)
* Max Inspiratory Positive Airway Pressure (IPAP) = 25 cm H2O
* Min Pressure Support (PS) = 2 cm H2O (cannot be adjusted)
* MaxPS = 8 cm H2O
* Bi-Flex setting of 3

The SmartCard is inserted into the device to provide the programmed therapy. Both the participant and CPAP therapist will be blinded to the therapy the SmartCard is programmed to provide. The other supplies necessary to use the therapy at home will also be provided to the participant (i.e. mask, tubing, humidifier, etc.).

The CPAP therapist will also provide the training necessary to use the device at home and provide a number to call in case the participant encounters any difficulty using the device at home.

Standardized Counseling to Optimize Adherence to Therapy

Counseling to optimize adherence to CPAP therapy will consist of:

1. The clinician will discuss complaints regarding CPAP therapy to identify potential contributors to poor adherence to therapy. The standardized counseling to optimize adherence includes the following measures to address patient complaints and concerns:

   Interface
   * Assure current mask is properly applied and headgear is properly adjusted.
   * Persistent mask leaks or mask discomfort, skin trauma, or skin irritation will be addressed first by verifying mask and headgear adjustment and mask sizing. An alternate mask can be used if the problems cannot be addressed by fit or adjustment interventions.
   * If mouth leaks are the primary concern and a nasal mask is being used, then a nasal/oral mask will be considered or a chin strap will be offered in combination with nasal mask use.

   Therapy Side Effects
   * All patients will have initially been placed on a CPAP device with heated humidification. For continued oro-pharyngeal dryness, nasal dryness, nasal congestion, or rhinitis, humidification will be increased. Saline nasal sprays, steroids, or decongestants can be prescribed, if needed.
   * Dyspnea on CPAP or claustrophobia will be addressed with counseling as needed.
   * Note: Reducing the prescribed pressure to improve adherence will not be considered at this time.
2. A standardized description of obstructive sleep apnea (OSA) and its risks will be reviewed with the participant, as well as the American Academy of Sleep Medicine Fact Sheet Drowsy Driving (see Appendix III).
3. A standardized description of the evidence regarding the benefits of positive pressure therapy to treat OSA will be reviewed with the participant.

Participants will be instructed to use the device as much as possible while they are sleeping and to also make sure they allow an adequate opportunity to sleep each night.

ELIGIBILITY:
Participants who meet the inclusion/exclusion criterion below and are willing to participate in the protocol when contacted will be enrolled into the study. Participants need to meet all of the following inclusion criterion below:

Inclusion Criterion:

1. Age 21-75
2. New Diagnosis of OSA with a baseline respiratory disturbance index (RDI) ≥ 15 events/hr of sleep determined by either full night or split night PSG
3. Able and willing to provide written informed consent
4. Able to follow study procedures
5. Sub-optimal PSG titration with at least 3 hours of attempted PAP titration (defined below): and deemed by their physician as a titration failure

Sub-optimal PSG titration: at least one of the following:

1. Poor sleep efficiency during titration period (sleep efficiency ≤ 70%) (participants may be on sleep medications as per standard lab CPAP protocol ) or;
2. Frequent arousals based on three seconds of alpha frequency on EEG (non periodic limb movement (PLM)-related) of 20 or greater per hour during the titration portion of the study or;
3. CPAP titration aborted due to participant's request (due to intolerance), or
4. Persistent sleep disruption despite therapeutic CPAP therapy and in the judgment of the reviewing physician, suggesting a low probability to CPAP adherence

Exclusion Criteria:

1. Participation in another interventional research study within the last 30 days
2. Major uncontrolled medical or psychiatric condition such as congestive heart failure, neuromuscular disease, renal failure etc.
3. Prior CPAP or Bi-Level PAP use (within last 2 years)
4. Chronic respiratory failure or insufficiency, moderate Chronic Obstructive Pulmonary Disease (COPD) (FEV1 < 60%), or any known condition of an elevation of arterial carbon dioxide levels while awake
5. Surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days
6. Presence of an untreated, diagnosable, non-OSA related sleep disorder (e.g. restless legs syndrome, insomnia, etc.)
7. Periodic Limb movement arousal index of 10 or greater.
8. Refusal to consider further interventions to standard CPAP to optimize positive pressure therapy (e.g. different mask than what was used in lab)
9. PAP therapy otherwise medically complicated or contraindicated such as those with a difficult to size or adjust interface (mask) resulting in facial pain, skin irritation or trauma, or excessive air leaks
10. Shift workers or people experiencing jet lag
11. Known history of alcohol and or drug abuse
12. Diagnosis of Complex Sleep Apnea, (appears to be classic obstructive or mixed sleep apnea, but exhibits disruptive central apneas and periodic breathing on CPAP) 11, 12 or persistent central apnea during diagnostic PSG.
13. Diagnosis of Attention Deficit Hyperactivity Disorder
14. Chronic Hypnotic use (nightly use for three months or less)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Powell, Ph.D., Principal Investigator — Philips Respironics
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinics, Rochester, Minnesota
  - Clayton Sleep Institute, St Louis, Missouri

REFERENCES:
- [Result] Powell ED, Gay PC, Ojile JM, Litinski M, Malhotra A. A pilot study assessing adherence to auto-bilevel following a poor initial encounter with CPAP. J Clin Sleep Med. 2012 Feb 15;8(1):43-7. doi: 10.5664/jcsm.1658. PMID 22334808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 patients completing clinical polysomnography (PSG) with CPAP was assessed for study eligibility and consented to study participation across 3 study sites.
Pre-assignment Details: 3 participants aborted their PSG during titration and were not considered for randomization into this trial. They were not included in the baseline demographic analysis.
Period: Overall Study
Arm/Group | Auto BiLevel Group | CPAP Group
Started | 26 | 22
Completed | 26 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 51 patients completing clinical polysomnography with CPAP was assessed for study eligibility and consented to study participation. In regards to meeting suboptimal titrationinclusion criteria, 3 patients aborted their titration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Auto BiLevel Group | CPAP Group | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.5) | 56.6 (9.8) | 55.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 20 | 16 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 20 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48
College Education Level [Count of Participants; unit: Participants] — Number of participants that were college educated.
  Participants | 16 | 12 | 28
BMI [Mean (Standard Deviation); unit: kilograms per meter squared] | 34.9 (6.5) | 31 (4.4) | 33.0 (5.9)
Nicotine Use [Count of Participants; unit: Participants] — Number of participants who use nicotine: cigarettes, chewing tobacco or nicotine pills on a daily basis.
  Participants | 5 | 5 | 10
Alcohol Use [Count of Participants; unit: Participants] — Count of participants who drink: wine, beer, or hard alcohol on a weekly basis.
  Participants | 13 | 11 | 24
ATU-A, Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Attitudes Toward Use A asks 5 questions about self-efficacy of using the CPAP. Participants answer on a scale of 1 to 5, 1 - completely disagree and 5 - completely agree. The range response is 5 to 25, with 5 being the least confident in their CPAP usage and 25 being the most confident.
  units on a scale | 20.4 (3.2) | 19 (4.7) | 19.6 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Group Compliance of the Auto Bilevel Group Compared to the CPAP Group Measured by Average Nightly Use.
Description: Compliance was compared between the AutoBiLevel Group and the CPAP group by measuring the average use per night over the study period.
Time Frame: 90 days
Population: One randomized participant discontinued the study early (auto-bilevel Group). One participant in the CPAP group used therapy the first night and failed for the remainder of the study but completed all study visits.
Measure: Mean (Standard Deviation); unit: minutes/night
Arm/Group | Auto BiLevel Group | CPAP Group
Number analyzed (Participants) | 25 | 21
minutes/night | 284.7 (110.9) | 255.1 (116.9)
Statistical Analysis 1: Comparison: Auto BiLevel Group vs CPAP Group; Pilot study, not powered for any endpoint; Test type: Other — Pilot study, not powered for any endpoint; p = 0.377, Chi-squared

2. Primary Outcome: Percentage of Group Compliance of the Auto Bilevel Group Compared to the CPAP Group
Description: Percentage of Group Compliance was compared between AutoBiLevel Group and the CPAP group by measuring proportion of adherent users over the treatment period. Patients with compliance of at least four hours will be classified as "compliant" and those with less than four hours will be classified as "non-compliant". The % of compliant patients will be calculated using the cumulative number of hours on therapy divided by the total number of days of the investigation for each subject.
Time Frame: 90 days
Population: as for outcome 1
Measure: Number; unit: percentage of compliant users
Arm/Group | Auto BiLevel Group | CPAP Group
Number analyzed (Participants) | 26 | 22
percentage of compliant users | 62 | 55
Statistical Analysis 1: Comparison: Auto BiLevel Group vs CPAP Group; Test type: Other — Pilot study, not powered for any endpoint; p = .624, Chi-squared

3. Secondary Outcome: Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale is an 8 item questionnaire that measures the general level of daytime sleepiness. Participants were asked what the chance is they would doze off or fall asleep during different routine daytime situations. The survey answers questions on a scale of 0 to 3- 0 being no chance and 3 being a high chance of dozing. The lowest score possible is a 0 and the highest score possible is a 24.
Time Frame: Assessed at Baseline, Day 30 and Day 90
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auto BiLevel Group | CPAP Group
Number analyzed (Participants) | 26 | 22
units on a scale
  Basline | 9.7 (3.9) | 8.2 (4.6)
  Day 30 | 8.2 (3.2) | 6.6 (4.6)
  Day 90 | 8.1 (3.8) | 6.9 (4.4)

4. Secondary Outcome: Fatigue Severity Scale
Description: The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Participants answer questions on a scale of 1-7, 1 being Strongly Disagree and 7 being Strongly Agree. The scores can range from 9-63. The higher the score the higher the fatigue.
Time Frame: Assessed at Baseline, Day 30 and Day 90
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auto BiLevel Group | CPAP Group
Number analyzed (Participants) | 26 | 22
units on a scale
  Baseline | 4.6 (1.4) | 3.9 (1.0)
  30 day | 4.0 (1.2) | 3.7 (1.2)
  90 day | 3.9 (0.9) | 3.4 (1.2)

5. Secondary Outcome: Functional Outcomes of Sleep Quality
Description: Functional Outcomes of Sleep Quality consists of 30 questions related to the effects of fatigue on daily activities, the instrument was designed to evaluate the respondent's quality of life as it relates to disorders of excessive sleepiness. Five domains of day-to-day life are examined: activity levels, vigilance, intimacy and sexual relationships, productivity, and social outcomes. The participants answer on a scale of 0-4: 0 -I don't do this activity for other reasons,1-Yes, extreme, 2-Yes, moderate, 3-Yes, a little, 4-No. Scores can range 0-120, the lower the score the more tired or sleepy the participant is.
Time Frame: Assessed at Baseline, Day 30 and Day 90
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auto BiLevel Group | CPAP Group
Number analyzed (Participants) | 26 | 22
units on a scale
  Baseline | 84.0 (20.9) | 91.4 (17.3)
  30 day | 97.5 (13.8) | 96.6 (16.6)
  90 day | 100.0 (11.3) | 100.1 (15.4)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Auto BiLevel Group | CPAP Group
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No